CLINICAL TRIAL: NCT01629004
Title: Increasing Uptake of Colorectal Cancer Screening in Ontario
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: 308-2010
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Colorectal Disorders
Keywords: colorectal cancer; screening; fecal occult blood testing; mailed invitation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-responders (Other): Non-responders to an initial mailed CRC screening invitation from their family physician.
  FOBT kit. Mailed invitation.
  Interventions: Other: FOBT kit; Other: Mailed invitation
- Recall patients (Other): Those who responded to the initial mailed CRC screening invitation and are now due for repeat screening (i.e., "recall" patients).
  FOBT kit. Mailed invitation.
  Interventions: Other: FOBT kit; Other: Mailed invitation

INTERVENTIONS:
Other: FOBT kit — Mailed FOBT kit with educational materials and mailed CRC screening invitation on behalf of family physician.
  Other Names: Mailed FOBT kit
Other: Mailed invitation — Mailed CRC screening invitation alone on behalf of family physician.
  Other Names: Mailed invitation alone

SUMMARY:
The investigators hope to determine whether the addition of an FOBT kit and educational materials to a second mailed invitation compared to a second mailed invitation alone increases use of appropriate screening tests (FOBT for average risk or colonoscopy if increased risk) by eligible persons within 6 months of the second mailing in: (1)Non-responders to an initial mailed CRC screening invitation from their family physician and, (2)Those who responded to the initial mailed CRC screening invitation and are due for repeat screening (i.e., "recall" patients). In addition, the investigators will also explore the impact of the investigators intervention in likely under-screened groups such as those living in more remote areas of the province and those with low socio-economic status as well as assessing the cost-effectiveness of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a mailed CRC screening invitation through the CCO Invitation Pilot project
* No OHIP record of completion of FOBT since initial mailing (Non-responders arm only)
* No OHIP of 'CRC Cancer Screening Exclusion' tracking code since initial mailing (Non-responders arm only)
* An OHIP record of completion of FOBT 6 months since initial mailing (Recall arm only)
* Negative result according to LRT or if not in LRT, no record of interval colonoscopy in CIRT or OHIP (Recall arm only)

Exclusion Criteria:

* Age greater than 74 years at time of mailing
* Interval diagnosis of colorectal cancer
* Interval colonoscopy or flexible sigmoidoscopy
* Interval departure from Pilot physician's practice
* Death
* Presently institutionalized
* Physician has declined participation in the study
* Interval record of repeat FOBT (Recall arm only)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5155 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Uptake of appropriate CRC screening | Within 6 months of the mailing
  The primary outcome will be the uptake of appropriate screening (FOBT testing or if there is a positive family history, of colonoscopy) within 6 months of the mailing as determined by from OHIP and CCO data.

SECONDARY OUTCOMES:
Uptake of lower gastrointestinal investigations | Within 12 months of the mailing
  The secondary outcome will be the uptake of lower gastrointestinal investigations (colonoscopy for an indication other than family history or colonoscopy done outside of CIRT, flexible sigmoidoscopy, barium enema) within 12 months, respectively, of the mailing as determined by the administrative data (CIRT, OHIP procedure or radiology code).

CONTACTS AND LOCATIONS:
Overall Officials: Jill Tinmouth, MD, Principal Investigator — Sunnybrook HSC
Locations (1):
- Sunnybrook HSC, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tinmouth J, Patel J, Austin PC, Baxter NN, Brouwers MC, Earle C, Levitt C, Lu Y, Mackinnon M, Paszat L, Rabeneck L. Increasing participation in colorectal cancer screening: results from a cluster randomized trial of directly mailed gFOBT kits to previous nonresponders. Int J Cancer. 2015 Mar 15;136(6):E697-703. doi: 10.1002/ijc.29191. Epub 2014 Sep 23. PMID 25195923